CLINICAL TRIAL: NCT01716091
Title: The Effect of Saline Irrigation in the Peritoneal Cavity at Cesarean Delivery on Maternal Morbidity and Gastrointestinal System Outcome
Brief Title: The Effect of Saline Irrigation in the Peritoneal Cavity at Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, T.C. Şişli Etfal E A H, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Other Study IDs: Aşıcıoğlu 02
Record Dates: First submitted 2012-10-22; First posted 2012-10-29 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Postoperative Enfectious Morbidity; Postoperative GİS Functionally Recovery
Keywords: focus of study is postoperative enfectious morbidity and postoperative GİS functionally recovery
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- saline irrigation: irrigation group:saline irrigation after uterine wall closed control group:no irrigation after uterine wall closed
  Interventions: Procedure: irrigation in the peritoneal cavity

INTERVENTIONS:
Procedure: irrigation in the peritoneal cavity — irrigation in the peritoneal cavity after uterine wall closed at cesarean

SUMMARY:
The investigators hypotheised that irrigating the abdominal cavity with saline at the time of cesarean delivery will increase Gastrointestinal System Disfunction without maternal infectious morbidity(especially febril morbidity).

ELIGIBILITY:
Inclusion Criteria:

1. Elective cesarean delivery
2. Gestational age greater 38 weeks

Exclusion Criteria:

1. chorioamnıonıtıs
2. type 1 diabetes mellitus
3. placenta previa and acreata
4. prior severe gastrointestional disease
5. emergency cesarean delivery

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all pregnant women between 18 years or older and who requıred cesarean delivery.
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
postoperative gastrointestinal system disturbance | postoperativeone weeks
  ıntraoperative and postoperative nausea,emesiz and requirement antıemetic drug

SECONDARY OUTCOMES:
postoperative febril morbidity | postoperative six weeks
  postoperative endometritis,febril morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Osman Aşıcıoğlu, M.D., Principal Investigator — T.C. Kanuni Sultan Süleyman Teaching Hospital
Locations (1):
- T.C. Kanuni Sultan Süleyman Teaching Hospital, Halkalı/İstanbul, Küçükçekmece, Turkey (Türkiye)